CLINICAL TRIAL: NCT06605300
Title: The Modulatory Effects of Oxytocin and Vasopressin on Delta-beta Cross-frequency Coupling
Brief Title: The Effects of Oxytocin and Vasopressin on Delta-beta Cross-frequency Coupling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Shuxia Yao, Associate Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-96
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: oxytocin; vasopressin; delta-beta coupling
MeSH Terms: conditions — Diabetes Insipidus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- oxytocin (Experimental): A single dose of 24 international units (IU) of oxytocin will be administered with 3 puffs of treatment to each nostril.
  Interventions: Drug: Intranasal Oxytocin (IN-OXT)
- vasopressin (Experimental): A single dose of 20 international units (IU) of vasopressin will be administered with 3 puffs of treatment to each nostril.
  Interventions: Drug: Intranasal Vasopressin (AVP)
- placebo (Placebo Comparator): A single dose of placebo will be administered with 3 puffs of treatment to each nostril.
  Interventions: Drug: Intranasal Placebo

INTERVENTIONS:
Drug: Intranasal Oxytocin (IN-OXT) — Subject assigned to receive intranasal administration of oxytocin (24 IU).
  Arms: oxytocin
Drug: Intranasal Vasopressin (AVP) — Subjects assigned to receive intranasal administration of vasopressin (20 IU).
  Arms: vasopressin
Drug: Intranasal Placebo — Subjects assigned to receive intranasal administration of placebo.
  Arms: placebo

SUMMARY:
The main aim of the study is to investigate whether intranasal oxytocin and vasopressin have effects on delta-beta cross-frequency coupling under resting-state and task conditions.

DETAILED DESCRIPTION:
A double-blinded, placebo-controlled, between-subject design is employed in this study. In a randomized order, a total of 120 healthy males and females are instructed to self-administer intranasal spray of oxytocin, vasopressin, or placebo. (1) 15-minute resting-state EEG data are collected 35 minutes after treatment. (2) Participants complete tasks including Stroop, GO/NOGO, and anxiety induction with behavioral (response time, accuracy, or rating) and EEG data being collected. Personality traits of subjects are assessed using validated Chinese version questionnaires including the Beck Depression Inventory (BDI-II), State-Trait Anxiety Inventory (STAI), Autism Spectrum Quotient (ASQ), and Adult ADHD Self-Report Scale (ASRS-v1.1). Participants are asked to complete Positive and Negative Affect Schedule (PANAS) when they just arrive, before resting state and after the tasks. Three blood samples (5 ml) are collected into 6 ml ETDA tubes when participants just arrive, before resting state recording and after all of the tasks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without past or current psychiatric or neurological disorders.

Exclusion Criteria:

* History of head injury.
* Pregnant,menstruating,taking oral contraceptives.
* Medical or psychiatric illness.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2024-10-02 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Resting-state EEG | 35-50 minutes after treatment administration.
  Participants are asked to sit comfortably and look at a white cross fixation against a black background on the computer monitor for 15 minutes with delta-beta cross-frequency coupling as a main index.
Behavioral indices in the tasks | 50-90 minutes after treatment administration.
  Reaction time and accuracy are recorded in the emotional Stroop and Go/Nogo tasks. For the anxiety induction task, participants are instructed to rate their anxiety levels using a 9-point Likert scale within 4 seconds (1 = not at all, 9 = very anxious).
Task-based EEG | 50-90 minutes after treatment administration.
  EEG data are recorded in the emotional Stroop, Go/Nogo, and anxiety induction tasks. Delta-beta cross-frequency coupling will be calculated to do statistical analyses.

SECONDARY OUTCOMES:
SCR in anxiety induction | 70-90 minutes after treatment administration.
  Skin Conductance Response (SCR) data are recorded in the anxiety induction task under safe and anxious conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Shuxia Yao, Dr, Principal Investigator — University of Electronic Science and Technology of China
Locations (2):
- China (2):
  - University of Electronic Science and Technology of China, Chengdu, Chengdu
  - University of Electronic Science and Technology of China (UESTC), Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No